CLINICAL TRIAL: NCT01852721
Title: Gender Differences in Response to the Mediterranean Diet-Part 2
Brief Title: Effects of the Mediterranean Diet on Cardiovascular Risk Profile in Men and Women (ALIMED)-Part 2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Laval University (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); Heart and Stroke Foundation of Canada (Other)
Responsible Party: Principal Investigator, Simone Lemieux, Professor, Laval University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2009-213 A1; MOP 84568 (Other Grant/Funding Number: Canadian Institutes of Health Research (MOP 84568)); 2007-180 (Other Grant/Funding Number: Heart and Stroke Foundation of Quebec (2007-180))
Record Dates: First submitted 2013-05-09; First posted 2013-05-14 (Estimated); Last update posted 2013-09-06 (Estimated); Status verified 2013-09

CONDITIONS: Cardiovascular Diseases
Keywords: Cardiovascular diseases; Nutritional intervention program; Self-Determination Theory; Motivational interviewing; Gender differences; Women; Men; Motivation; Dietary intakes; Mediterranean diet; Eating behaviors; Lipid profile
MeSH Terms: conditions — Cardiovascular Diseases; Multiple Endocrine Neoplasia Type 1; Feeding Behavior | interventions — Diet, Mediterranean

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Men and Mediterranean diet (Experimental): The 12-week nutritional education program will include 3 group sessions with 8-12 participants per group, 3 individual counseling sessions, and 4 telephone interviews. The registered dietitian will encourage participants to make their own decision about dietary changes while promoting their autonomy and competence, and will accept participants' choices, avoiding pressuring them to perform a specific change.
  Interventions: Behavioral: Experimental: Men and Mediterranean diet
- Women and Mediterranean diet (Experimental): The 12-week nutritional education program will include 3 group sessions with 8-12 participants per group, 3 individual counseling sessions, and 4 telephone interviews. The registered dietitian will encourage participants to make their own decision about dietary changes while promoting their autonomy and competence, and will accept participants' choices, avoiding pressuring them to perform a specific change.
  Interventions: Behavioral: Experimental: Women and Mediterranean diet

INTERVENTIONS:
Behavioral: Experimental: Men and Mediterranean diet — The 12-week nutritional education program will include 3 group sessions with 8-12 participants per group. During the 1st group session, the registered dietitian (RD) will explain the major principles of the Mediterranean diet (MedDiet) and related heath benefits. At week 4, subjects will be invited to a Mediterranean cooking lesson. At week 8, the group session will address barriers and difficulties in adhering to the recommendations. Individual sessions will take place at weeks 1, 5 and 10 in order to evaluate the dietary changes and to select further individualized objectives for increasing the adherence to the MedDiet. The RD will encourage participants to make their own decision about changes while promoting their autonomy and competence. Qualitative 24-h recalls will be performed by telephone at weeks 3, 6, 9 and 12 to reinforce key principles of the MedDiet. No further contact with the RD will be offered during the follow-up period.
  Arms: Men and Mediterranean diet
Behavioral: Experimental: Women and Mediterranean diet — Women are assigned to the same intervention than men in order to compare men and women adherence to the Mediterranean diet.
  Arms: Women and Mediterranean diet

SUMMARY:
The purpose of this study is to document differences between men and women (referred here as gender differences) in diet adherence and in changes in specific dietary intakes and energy density in response to a 12-week nutritional education program promoting the Mediterranean diet in both the short term (immediately after the end of the intervention) and longer term (3 and 6 months after the end of the intervention). The investigators hypothesize that both in the short and the longer term, women will have a better adherence to recommendations promoting the Mediterranean diet than men namely because of higher self-determination.

DETAILED DESCRIPTION:
Among the few studies that have addressed gender differences in response to a nutritional program promoting the Mediterranean diet, none has used a theoretical model of dietary adherence. Accordingly, the Self-Determination Theory suggests that the different behavioral types of regulation are associated with one of the three forms of motivation which are intrinsic motivation, extrinsic motivation and amotivation. The use of the Self-Determination Theory as a theoretical model of adherence will provide original data on the potential contribution of self-determination to gender differences in adherence to an intervention promoting the Mediterranean diet. The purpose of this study is to document gender differences between men and women in diet adherence and in changes in specific dietary intakes and energy density in response to a 12-week nutritional education program promoting the Mediterranean diet in both the short term (immediately after the end of the intervention) and longer term (3 and 6 months after the end of the intervention). Considering that previous studies have shown that women were more likely than men to take action to improve eating habits, rated higher their knowledge of nutrition than men and also indicated that they read product labels more frequently than men, we hypothesize that both in the short and the longer term, women will have a better adherence to recommendations promoting the Mediterranean diet than men namely because of higher self-determination. Data will be collected before and after the 12-week nutritional education program, as well as 3 and 6 months after the end of the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Men and premenopausal women from de Quebec City metropolitan area.
* Involved in food purchases and/or meal preparation
* Stable body weight (+/- 2.5 kg) for at least 3 months before the beginning of the study
* Slightly elevated LDL-cholesterol concentrations (≥ 3.0 mM) or total cholesterol to HDL-C ratio ≥ 5.0
* At least one of the four following factors of the metabolic syndrome:

  1. Triglycerides ≥ 1.7 mM;
  2. Fasting glucose between 6.1 and 6.9 mM;
  3. Blood pressure concentrations ≥ 130 / 85 mm Hg;
  4. Waist circumference > 94 cm in men and > 80 cm in women

Exclusion Criteria:

* Smokers
* Alcoholism problem
* Pregnancy
* Cardiovascular and endocrinal diseases
* Medication that could affect dependent variables measured (namely lipid-lowering, hypoglycemic, insulin sensitizers and antihypertensive medication)
* Food allergies/aversions
* Mediterranean score > 29

Ages: 25 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 123 (Actual)
Dates: Start 2010-03; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Diet adherence | At baseline (t=0) and immediately after the 12-week intervention (t=3 mo) as well as 3 (t=6 mo) and 6 months (t= 9 mo) after the end of the intervention.
  A Mediterranean score will be used to measure diet adherence. As described by Dansinger et al, we will use a 10-point score to describe the degree to which each subject achieves the specified dietary target vs baseline intakes. The target would be a perfect Mediterranean score of 44. For example, a subject with a Med Score of 20 at baseline and of 30 at t=12 weeks will therefore have an adherence score at t=12 weeks of : (20 - 30) / (20 - 44) =0.42 or 4.2 on a scale of 10.

SECONDARY OUTCOMES:
Dietary intakes | At baseline (t=0) and immediately after the 12-week intervention (t=3mo) as well as 3 (t=6 mo) and 6 months (t= 9 mo) after the end of the intervention.
  A 30-min Food Frequency Questionnaire (FFQ) will be administered face-to-face by a Registered Dietitian. A Mediterranean score will be derived from the FFQ. The Mediterranean score could therefore vary between 0 and 44 points.
  A 3-day weighed food record will be completed in order to derive a precise measurement of energy density.
Eating behaviors | At baseline (t=0) and immediately after the 12-week intervention (t=3 mo) as well as 3 (t=6 mo) and 6 months (t= 9 mo) after the end of the intervention.
  Cognitive dietary restraint, disinhibition, and susceptibility to hunger.
Anthropometric and metabolic parameters | At baseline (t=0) and immediately after the 12-week intervention (t=3 mo) as well as 3 (t=6 mo) and 6 months (t= 9 mo) after the end of the intervention.
  Anthropometric variables (height, weight, waist and hip circumferences) according to standardized procedures and basic lipid profile, fasting glycemia and insulinemia as well as blood pressure will be measured.
Physical activity level | At baseline (t=0) and immediately after the 12-week intervention (t=3 mo) as well as 3 (t=6 mo) and 6 months (t= 9 mo) after the end of the intervention.
  A validated 3-day physical activity record (two weekdays and one weekend day).
Global motivational variables | At baseline (t=0).
  Self-Determination Scale. Basic Psychological Needs Scale.
Motivational variables in a nutrition context | At baseline (t=0) and immediately after the 12-week intervention (t=3 mo) as well as 3 (t=6 mo) and 6 months (t= 9 mo) after the end of the intervention.
  Regulation of Eating Behaviors Scale.
Quality of life | At baseline (t=0) and immediately after the 12-week intervention (t=3 mo) as well as 3 (t=6 mo) and 6 months (t= 9 mo) after the end of the intervention.
  SF-36.
Health-Care Climate | After the end of the 12-week intervention (t=3 mo).
  Health-Care Climate Questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Simone Lemieux, Ph.D., Dt.P, Principal Investigator — Department of food sciences and nutrition / Institute of Nutraceutical and Functional Foods (INAF), Laval University
Locations (1):
- Institute of Nutraceuticals and Functional Foods (INAF), Laval University, Québec, Quebec, Canada

REFERENCES:
- [Derived] Leblanc V, Begin C, Hudon AM, Royer MM, Corneau L, Dodin S, Lemieux S. Gender differences in the long-term effects of a nutritional intervention program promoting the Mediterranean diet: changes in dietary intakes, eating behaviors, anthropometric and metabolic variables. Nutr J. 2014 Nov 22;13:107. doi: 10.1186/1475-2891-13-107. PMID 25416917